CLINICAL TRIAL: NCT04686825
Title: A Randomized, Open-label, Single-dose, 4-way Crossover Phase 1 Study to Evaluate the Food Effect on Pharmacokinetics of DA-8010 After a Single Administration of DA-8010 2.5 mg or 5 mg in Healthy Subjects
Brief Title: The Food Effect on Pharmacokinetics of DA-8010 After a Single Administration of DA-8010 2.5 mg or 5 mg in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DA8010_DIF_I
Record Dates: First submitted 2020-12-23; First posted 2020-12-29 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-01

CONDITIONS: Healthy
MeSH Terms: interventions — DA-8010

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- T1 (Experimental): DA-8010 2.5 mg (Fasting)
  Interventions: Drug: DA-8010 2.5mg (Fasting)
- T2 (Experimental): DA-8010 2.5 mg (Fed)
  Interventions: Drug: DA-8010 2.5mg (Fed)
- T3 (Experimental): DA-8010 5 mg (Fasting)
  Interventions: Drug: DA-8010 5mg (Fasting)
- T4 (Experimental): DA-8010 5 mg (Fed)
  Interventions: Drug: DA-8010 5mg (Fed)

INTERVENTIONS:
Drug: DA-8010 2.5mg (Fasting) — Test drug l : DA-8010 2.5mg (Fasting)
  Arms: T1
Drug: DA-8010 2.5mg (Fed) — Test drug ll : DA-8010 2.5mg (Fed)
  Arms: T2
Drug: DA-8010 5mg (Fasting) — Test drug llI : DA-8010 5mg (Fasting)
  Arms: T3
Drug: DA-8010 5mg (Fed) — Test drug lV : DA-8010 5mg (Fed)
  Arms: T4

SUMMARY:
This is a randomized, open-label, single-dose, 4-way crossover phase 1 study to evaluate the food effect on pharmacokinetics of DA-8010 after a single administration of DA-8010 2.5 mg or 5 mg under fasting and fed states in healthy male and female subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteer 19 years to 50 years
* Body weight in the range of 45.0 to 90.0 kg and body mass index in the range of 18 to 30kg/m2
* The subjects personally signed and dated informed consent document after informed of all patient aspects of the study, fully understanding and determined spontaneously to participate
* The subjects who are judged appropriate to participate this clinical trial according to the physical examination, routine laboratory examination and questionnaire

Exclusion Criteria:

* Subject with serious active hepatobiliary (severe hepatic failure, etc.), renal(severe renal impairment, etc.), neurologic, immunologic, respiratory, digestive, endocrine, hematologic, cardiovascular(heart failure, Torsades de pointes, etc), urologic, psychological disease or history of such disease
* Subject Hypersensitive to any of the IP components or other drug components(Aspirin, Antibiotics, etc.)
* Subject with gastrointestinal disease (peptic ulcer, gastritis, gastrospasm, gastroesophageal reflux disease, Crohn's disease, etc.) or history of such disease/surgery (excluding simple appendic surgery, hernia surgery, hemorrhoid surgery)
* Subject who have blood pressure < 90 mmHg or >150 mmHg as systolic or <60 mmHg or >100 mmHg as diastolic
* Subject who have history of drug abuse or Positive in Urine drug screen test
* Subject who are Positivie in Alcohol breath test on screening
* Subject who have ETC drug or oriental medicine 2 weeks prior to IP administration or OTC drug or health functional food or vitamins 1 week prior to IP administration
* Subject who have taken a drug that induces or inhibits the drug metabolic enzyme (e.g., barbital) within 30 days prior to IP administration
* Subject who have participated in other clinical trials within 6 months prior to the first administration of the IP
* Subject who have had whole blood transfusion within 2 months or the apheresis within 2 weeks prior to the first administration of the IP
* Subject with a history of regular alcohol intake(>21 units/week , 1 unit = 10 g of pure alcohol) or who are unable to quit alcohol from 3 days prior to the first administration of the IP until out of hospital
* Smoker(excluding who quit smoking 3 months before this clinical trial) or subject who are unable to quit smoking from 3 days prior to first administration of the IP until out of hospital
* Subject who are unable to quit food containing grapefruit from 3 days before first administration of the IP until out of hospital
* Subject who regularly intake caffeine(> 5 units/day) or who are unable to quit caffeine/food containing caffeine from 3 days before first administration of the IP until out of hospital
* Subject with unusual eating habits (continuous vegetarian diet, etc.) or who are unable to consume the entire diet provided in this clinical trial
* Subject who are positive in pregnancy test or pregnant or Lactating women
* Subject who do not agree to exclude the possibility of pregnancy using the contraception from the date of the first administration of the IP until the 4 weeks after the last administration.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2021-02-17 (Actual); Study Completion 2021-03-11 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 0~48hours
  PK parameter
Area under the plasma concentration versus time curve (AUClast) | 0~48hours
  PK parameter

CONTACTS AND LOCATIONS:
Overall Officials: Seung Hwan Lee, PhD, Principal Investigator — SNUH Clinical Pharmacololgy and Therapeutics
Locations (1):
- Seoul National University Hospital, Soeul, South Korea